CLINICAL TRIAL: NCT00914446
Title: Identification of Protective and Worsening Steatohepatitis (NASH) Factors by Microarray in Morbid Obesity Patients
Brief Title: Identification of Protective and Worsening Steatohepatitis (NASH) Factors
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Département de la Recherche Clinique - Mme MALERBA, Centre Hospitalier Universitaire de Nice
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 07-APR-05
Record Dates: First submitted 2009-04-15; First posted 2009-06-05 (Estimated); Last update posted 2009-06-05 (Estimated); Status verified 2009-06

CONDITIONS: Morbid Obesity; Steatohepatitis; Steatosis
Keywords: Steatohepatitis
MeSH Terms: conditions — Obesity, Morbid; Fatty Liver

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- morbid obese subject (Other)
  Interventions: Procedure: hepatic biopsies
- overweight and NASH subjects (Other)
  Interventions: Procedure: hepatic biopsies
- control subjects (Other)
  Interventions: Procedure: hepatic biopsies

INTERVENTIONS:
Procedure: hepatic biopsies — hepatic biopsies

SUMMARY:
The main aim of this work will be to identify a profile of gene expression by microarray in the liver which might allow to differentiate obese subjects having a normal liver from those with steatohepatitis or steatosis.

DETAILED DESCRIPTION:
Recent epidemiological studies in France showed a strong prevalence of obesity (12,4%) and its strong increase during the 20 last years. Among the multiple complications related to obesity, the hepatic complications (steatosis and steatohepatitis (NASH)) are among most frequent. Our recent work showed that the adipose tissue, following the example of hepatic tissue also expressed CRP, the hepcidin and the IL-6 on a gene and protein level. We also noticed that 5% of our patients in spite of their obesity presented a normal liver without steatosis.

The main aim of this work will be to identify a profile of gene expression by microarray in the liver which might allow to differentiate the obese subjects having a normal liver from those with steatohepatitis or steatosis. The gene studies will be carried out initially in morbid obese subjects without diabetes (women, index of body mass > 40 kg/m2). We will select a sample of 10 patients having a normal liver, 10 patients having a NASH and 10 patients having a simple steatosis. These gene studies will be carried out in the liver and visceral adipose tissue from these same patients which will make possible to evaluate the interrelationship between the liver and the adipose tissue. We will also include 10 patients having an overweight and a NASH (study only on liver biopsy). The livers controls (10) will be provided from the department of surgery of Pr Jean Gugenheim and are practically all available. They are "healthy" tissue near hepatic benign tumors. Commercial ARN (Biosciences, Stratagene) will be also used. After identification of these profiles of gene expression in a restricted number of patients, we will validate these profiles of gene expression in a more significant number of patients (30 to 45 patients having a NASH compared with 30 to 45 patients having a simple steatosis).

The secondary objectives will be:

To compare the profile of gene expression between the liver and the adipose visceral and subcutaneous tissue from the morbid obese subjects After the identification of a group of genes of interest whose expression is modified in a small number of patients having a NASH, we continue our study with a more restricted number of genes.

* To validate in a more significant number of patients the modifications of expression of these genes by an approach by real-time PCR
* To determine the site of expression of these factors in the liver or adipose tissue by immunohistochemic analysis
* To determine the rate of expression of these factors in the liver or adipose tissue by biochemical analysis (Western blot)
* A serum dosage could finally be carried out to determine if the serum proteins could constitute a predictive index of the NASH or steatosis.

We will use the series of obese patients from the CHU of Nice whose a surgical approach of obesity was programmed. Preoperative explorations include clinico-biological assessments. During the intervention, the liver and adipose tissue biopsies will be systematically realized for research. We will also use the hepatic biopsies carried out among patients having an overweight and a NASH.

The feasibility of the work does not pose any problem. The department of surgery carries out 10 surgeries of obesity per month. We already have a series of 280 patients. We must include 150 patients in order to be able to obtain sufficiently patients with normal liver. For the other patients, we will use the tissue bank which is already carried out and the patients already gave the consent. Finally we must constitute a liver tissue bank for patients having an overweight. All these fundamental techniques are controlled within team from INSERM U 568 Awaited results: We could by this strategy select protective and worsening factors of steatohepatitis (NASH) which will be able to lead to identify predictive biological markers of the lesions of steatohepatitis and thus to identify patients at risk for the hepatic lesions. These factors could also serve as future therapeutic targets.

ELIGIBILITY:
Inclusion Criteria for morbid obese subjects without diabetes:

* 18-60 years old, male or female
* Body mass index > 40 kg/m2
* Obesity surgery required
* Alcohol consumption < 20g per day
* Affiliation to national French health insurance
* Consent agreement

Exclusion criteria:

* Hepatitis B, C, HIV
* Pregnant or breast-feeding woman.
* Inability to sign informed consent
* Patient with regulatory authority patient gold private freedom
* Hémochromatosis
* Toxic Hepatitis
* Alpha-1-anti-trypsin Deficiency
* Wilson disease
* Auto-immune hepatitis
* Drug Hepatitis
* Orlistat

Inclusion criteria for controls subjects:

* Subjects of the 2 sexes of 18-60 years old
* Patients with normal body mass index between 20-25 kg/m2
* Patients profiting from hepatectomy for benign tumors like adenoma or bulky tumor hepatic biliary cyst or from a repair of the abdominal wall
* Subjects affiliated to a mode of social security
* Patient having signed the enlightened consent
* The private subjects from freedom and the major subjects under supervision will be excluded

Inclusion criteria for overweight and NASH subjects:

* Subjects of the 2 sexes of 18-60 years old
* Patients with body mass index > 25 kg/m2
* Alcohol Consumption < 20 g/j
* Patient having a NASH in the hepatic biopsy
* Subjects affiliated to a mode of social security
* Patient having signed the enlightened consent

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 150 (Estimated)
Dates: Start 2008-04; Primary Completion 2009-12 (Estimated); Study Completion 2010-04 (Estimated)

PRIMARY OUTCOMES:
Anatomopathologic study of the hepatic biopsies. | one day

SECONDARY OUTCOMES:
Seek protective and worsening factors by "microarray" | one day
Quantitative analyses of genes of interest in the liver and and visceral adipose tissue | one day
Immunohistochemical analyses | one day
Biochemical analyses | one day
Serum dosage of protein of interest | one day

CONTACTS AND LOCATIONS:
Overall Officials: ALBERT TRAN, Ph D, Principal Investigator — Centre Hospitalier Universitaire de Nice
Locations (1):
- CHU de Nice Hôpital de l'Archet, Nice, NICE, France